CLINICAL TRIAL: NCT07043790
Title: Radical Cystectomy Versus Tri-Modal Therapy for Treatment of cT2N0M0 Urinary Bladder Transitional Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Himdan Abdelhameed, Assistant Lecturer of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD 183/2022
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Transitional Cell Bladder Cancer; Cystectomy; Radiation
MeSH Terms: interventions — Cystectomy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial comparing radical cystectomy and trimodal therapy, included adult patients with cT2N0M0 muscle invasive localized urinary bladder TCC presented to our urology clinic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical Cystectomy group (Active Comparator): Gtoup A : Radical cystectomy group Radical cystectomy included surgical removal of the bladder, adjacent organs, and regional lymph nodes. In males, it included removal of urinary bladder, prostate, and seminal vesicles whereas in females, it included removal of urinary bladder and reproductive organs (ovaries, fallopian tubes, uterus, and anterior vagina).
  Standard pelvic lymph node dissection was performed to all patients in this group.
  Interventions: Other: Radical cystectomy with pelvic lymphadenectomy
- Trimodal therapy group (Active Comparator): Group B : trimodal therapy group
  the patients underwent maximal TURBT, where as much tumor as possible was completely resected using bipolar resectoscope. The goal was to remove all visible tumor including the underlying muscle layer and tumor edges.
  This was followed by radio-sensitizing chemotherapy and radiotherapy..
  Chemotherapy consisted of weekly administration of iv infusion of cisplatin (40mg/m2).
  Radiotherapy delivered as EBRT aimed at delivering approximately 44- 46 Gy to the urinary bladder and pelvic lymphnodes.followed by additional boost to the bladder 54 GY and a final boost to the tumor 64-65 GY
  Interventions: Radiation: Trimodal therapy

INTERVENTIONS:
Other: Radical cystectomy with pelvic lymphadenectomy — Gtoup A : Radical cystectomy group Radical cystectomy included surgical removal of the bladder, adjacent organs, and regional lymph nodes. In males, it included removal of urinary bladder, prostate, and seminal vesicles whereas in females, it included removal of urinary bladder and reproductive organs (ovaries, fallopian tubes, uterus, and anterior vagina).
  Standard pelvic lymph node dissection was performed to all patients in this group.
  Arms: Radical Cystectomy group
Radiation: Trimodal therapy — Group B : trimodal therapy group
  the patients underwent maximal TURBT, where as much tumor as possible was completely resected using bipolar resectoscope. The goal was to remove all visible tumor including the underlying muscle layer and tumor edges.
  This was followed by radio-sensitizing chemotherapy and radiotherapy..
  Chemotherapy consisted of weekly administration of iv infusion of cisplatin (40mg/m2).
  Radiotherapy delivered as EBRT aimed at delivering approximately 44- 46 Gy to the urinary bladder and pelvic lymphnodes.followed by additional boost to the bladder 54 GY and a final boost to the tumor 64-65 GY
  Arms: Trimodal therapy group

SUMMARY:
the aim of this study is to compare the oncological outcome of trimodal therapy with bladder preservation using maximal resection with chemoradiation versus the standard radical cystectomy for muscle invasive transitional cell carcinoma of urinary bladder.

DETAILED DESCRIPTION:
Bladder cancer is the 9th most common cancer in the world, accounting for approximately 5-8% of all male cancers which makes it the 4th most common cancer in men and accounts for approximately 2% of female cancers making it the 8th most common cancer among women .

Bladder cancer is the 2nd most common urogenital cancer; thus, it is considered a very frequent disease to deal with in urological practice .

The urinary bladder is lined internally with transitional epithelial cells (urothelium), followed by lamina propria which is formed of connective tissue supporting the overlying urothelium, then muscularis propria (detrusor muscle) followed by an outer layer called serosa .

Bladder cancer is usually presented by gross or microscopic hematuria (85-90%), it may be associated with irritative symptoms, especially in the presence of carcinoma in situ.

In advanced disease, the patient may complain of bone pain, loin pain, pain radiating to the buttocks and thighs, or even renal impairment due to obstruction of both lower ureters.

Diagnosis and staging of bladder cancer are multimodal approaches done through a combination of clinical, radiological, and histopathological means.

Magnetic resonant imaging MRI lacks ionizing radiation, so it is considered a safe way to investigate a patient with cancer bladder before, during, or following up the treatment to determine its response .

Diagnostic cystoscopy is the only definitive diagnostic tool through histopathological examination of the resected tissues. Proper sampling should include the underlying muscularis propria. Transurethral resection of bladder tumor (TURBT) can miss proper muscle layer sampling in 25% of invasive cancer leading to under-staging. TURBT depends on the surgeon's experience, so the tumor-free rate varies widely .

Differentiation between non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC) is a cornerstone in the treatment plans. Treatment methods aim at preserving the quality of life and reduce stage progression. The usual conservative approach in MIBC is a trimodal treatment (TMT). It consists of a transurethral resection of the bladder tumor (TURBT) as complete as possible, followed by concomitant radiotherapy (RT) and chemotherapy (CT). Response to radiotherapy and chemotherapy is then assessed by cystoscopy and biopsies. Planned surgery is proposed to non-responders and additional chemotherapy and RT with careful regular endoscopic examination is performed in responders .

Except for the incomplete selective bladder preservation against radical excision (SPARE) trial, there is no large and meaningful randomized trial comparing radical cystectomy and TMT .

ELIGIBILITY:
Inclusion Criteria:

* Adults of any gender, aged 18 years or older.
* Histologically confirmed urothelial (transitional cell) carcinoma (TCC) of the urinary bladder, clinical stage T2N0M0, diagnosed through:

  * Imaging (CT or MRI).
  * Cystoscopy.
  * Biopsy and histopathological examination of the tumor.

Exclusion Criteria:

* Evidence of significant nodal involvement on imaging.
* Presence of carcinoma in situ (CIS).
* Hydronephrosis attributed to the bladder tumor.
* Non-TCC histology of bladder cancer.
* TCC with atypical histological variants including:

  * Micropapillary,
  * Plasmacytoid,
  * Anaplastic, or
  * Sarcomatoid variants.
* High-grade non-muscle invasive bladder cancer (NMIBC).
* Patients unfit for surgery.
* Patients unfit for chemotherapy or radiotherapy.
* Refusal to undergo randomization.
* Prior chemotherapy or radiotherapy for bladder cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
Disease free survival | 3 years
Cancer specific survival | 3 years

SECONDARY OUTCOMES:
Complications of intervention | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Lotfy Ghazy, Lecturer of Urology, Study Director — Ain Shams University
Locations (1):
- AIn shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Result] Kulkarni GS, Black PC, Sridhar SS, Kapoor A, Zlotta AR, Shayegan B, Rendon RA, Chung P, van der Kwast T, Alimohamed N, Fradet Y, Kassouf W. Canadian Urological Association guideline: Muscle-invasive bladder cancer. Can Urol Assoc J. 2019 Aug;13(8):230-238. doi: 10.5489/cuaj.5902. No abstract available. PMID 30763236
- [Result] Imai S, Yamada T, Kasashi K, Niinuma Y, Kobayashi M, Iseki K. Construction of a risk prediction model of vancomycin-associated nephrotoxicity to be used at the time of initial therapeutic drug monitoring: A data mining analysis using a decision tree model. J Eval Clin Pract. 2019 Feb;25(1):163-170. doi: 10.1111/jep.13039. Epub 2018 Oct 2. PMID 30280456
- [Result] Ritch CR, Balise R, Prakash NS, Alonzo D, Almengo K, Alameddine M, Venkatramani V, Punnen S, Parekh DJ, Gonzalgo ML. Propensity matched comparative analysis of survival following chemoradiation or radical cystectomy for muscle-invasive bladder cancer. BJU Int. 2018 May;121(5):745-751. doi: 10.1111/bju.14109. Epub 2018 Jan 22. PMID 29281848
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30280456/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30763236/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT07043790/Prot_SAP_000.pdf